CLINICAL TRIAL: NCT06140433
Title: Vital Signs Camera Study
Acronym: VSC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philips Clinical & Medical Affairs Global (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: IPS-200169-VSCstudy
Record Dates: First submitted 2023-10-11; First posted 2023-11-20 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Respiration Rate; Heart Rate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VSC-MEDlib (Other): SaMD: Data collection study. Software to be applied after data collection.
  Interventions: Device: VSC-MEDlib

INTERVENTIONS:
Device: VSC-MEDlib — VSC-MEDlib will be used for post-processing

SUMMARY:
This study is a single center, prospective clinical investigation which is balanced for gender, age, Body Mass Index (BMI) and skin color. Simultaneous measurements of PR and RR on study participants will be collected in conditions described in IFU and various suboptimal conditions. The study participants will be recorded with the VSC demo app (together with a compatible camera and computing hardware) and reference devices. PR and RR data to be collected by the VSC demo app, will be post-processed after the clinical investigation and compared with the reference devices. Persons who are willing to participate will be asked to provide their consent.

Primary objective:

• To assess the clinical safety and effectiveness of Pulse Rate (PR) and Respiration Rate (RR) measured with the VSC-MEDlib within the intended use compared to the gold-standard reference devices.

Exploratory objective:

• To assess the clinical safety and effectiveness of Pulse Rate and Respiration Rate measured with the VSC-MEDlib during suboptimal circumstances (outside the scope of the intended use), compared to the gold-standard reference devices.

ELIGIBILITY:
Inclusion Criteria:

* Persons with ASA I or II classification
* Adult population (age >18 years old)
* BMI ≥ 18 - ≤ 40 kg/m2
* Able to intensively exercise for 10 minutes
* Persons willing to give informed consent
* Willingness to have vital signs measured by a medical mobile application
* Willingness to follow study protocol (e.g., put on sunglasses, facial make-up, medical face-mask and sitting still up to 2 minutes)

Exclusion Criteria:

* Vulnerable populations (e.g., age <18 years old, not able to consent by themselves, or immunecompromised or pregnant women)
* Cardiac arrhythmias (e.g., Atrial Fibrillation, Supraventricular Tachycardia, Ventricular arrhythmia, regular ectopic beats)
* Persons present signs of infection
* Participant has known allergic reactions to make-up and/or make-up remover
* Persons with positive COVID 19 test in last 14 days
* Participant who exhibit irregular or excessive movement such as tremors, tics, shaking and/or shivering
* Participant is Philips employee or their family members residing with this Philips employee.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2024-02-02 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-03-15 (Actual)

PRIMARY OUTCOMES:
Clinical safety and effectiveness VSC-MEDlib according to IFU | 2 hours
  Clinical safety and effectiveness of the non-invasive and contactless measurement RR by the VSC-MEDlib within the intended use.
Clinical safety and effectiveness VSC-MEDlib according to IFU | 2 hours
  Clinical safety and effectiveness of the non-invasive and contactless measurement of PR by the VSC-MEDlib within the intended use.

OTHER OUTCOMES:
Clinical safety and effectiveness VSC-MEDlib during suboptimal conditions | 2 hours
  Safety and clinical effectiveness during suboptimal conditions, in RMSE, availability, and precision of the non-invasive and contactless measurement of RR by the VSCMEDlib.
Clinical safety and effectiveness VSC-MEDlib during suboptimal conditions | 2 hours
  Safety and clinical effectiveness during suboptimal conditions, in RMSE, availability, and precision of the non-invasive and contactless measurement of PR by the VSCMEDlib.

CONTACTS AND LOCATIONS:
Overall Officials: Murk Westerterp, Study Director — Integrated Technology Solutions
Locations (1):
- Philips, Eindhoven, North Brabant, Netherlands

IPD SHARING:
Plan to Share IPD: No